CLINICAL TRIAL: NCT01340508
Title: A Phase II Trial of Preoperative Concurrent Chemotherapy and (IMRT) in Locally Advanced Rectal Cancer
Brief Title: Preoperative Concurrent Chemotherapy and Intensity Modulated Radiotherapy (IMRT) in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Dr Jeremy Tey, National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B/09/377
Record Dates: First submitted 2011-04-18; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Rectal Cancers.
Keywords: Pathological complete response; Intensity modulated radiotherapy; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensity modulated Radiotherapy (Experimental): Intensity modulated radiotherapy, dose escalation, rectal cancer, volumetric modulated arc therapy
  Interventions: Radiation: Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy — Intensity modulated radiotherapy to a dose of 55Gy in 25 fractions
  Other Names: Intensity modulated radiotherapy. Dose escalation.

SUMMARY:
The hypothesis of this study is that dose escalated intensity modulated radiotherapy (IMRT) to a dose of 55Gy in 25# to primary rectal tumor concurrent with oral capecitabine results in an improved pathological response rate from 8% (German trial) to 25%.

DETAILED DESCRIPTION:
This study aims to look at whether radiation dose escalation with intensity modulated radiotherapy can increase the rates of pathological complete response in patients with locally advanced rectal cancer treated with neoadjuvant chemoradiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of adenocarcinoma of the rectum
* Clinically determined to be stage T3 or T4,N0-N2, and M0 -staged by MRI or transrectal ultrasound of the rectum
* Patients who are medically operable and who have resectable adenocarcinoma of the rectum at least <15cm from the anal verge
* Adequate liver/renal and haematological function.
* Eastern Cooperative Oncology Group (ECOG) performance 0-2
* Age ≥ 18 years
* Full blood count obtained within 2 weeks prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Haemoglobin ≥ 8.0 g/dl
* Serum creatinine within normal institutional limits or creatinine clearance ≥ 50 ml/min
* Bilirubin within normal institutional limits
* AST and ALT < 2.5 x the IULN
* Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years

* Prior systemic chemotherapy for colorectal cancer; note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 12 months
  * Transmural myocardial infarction within the last 6 months
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol.
  * Evidence of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
  * Known, existing uncontrolled coagulopathy. Patients on therapeutic anticoagulation may be enrolled provided that they have been clinically stable on anti-coagulation for at least 2 weeks.
  * Major surgery within 28 days of study enrollment (other than diverting colostomy)
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Prior allergic reaction to capecitabine
* Any evidence of distant metastases (M1)
* A synchronous primary colon carcinoma
* Extension of malignant disease into the anal canal
* Lack of physical integrity of the gastrointestinal tract (i.e., severe Crohn's disease that results in
* malabsorption; significant bowel resection that would make one concerned about the absorption of capecitabine) or malabsorption syndrome that would preclude feasibility of oral chemotherapy (capecitabine)
* Participation in any investigational drug study within 28 days of study enrollment

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rates | 8 weeks post chemoradiotherapy
  Pathogical complete response rate 8 weeks post chemoradiotherapy at surgery according to Ryan's classification

SECONDARY OUTCOMES:
Toxicity | 2 years
  Toxicity including anorexia, nausea, vomiting, diarrhoea, dermatitis, proctitis, urinary frequency/urgency as per common toxicity criteria v3.0
Disease Free survival | 2 years
  Time from study entry to disease recurrence or death
Downstaging rates | 8 weeks after chemoradiotherapy
  percentage of patients who achieve downstaging 8 weeks post chemoradiotherapy at surgery according to TNM classification
Sphincter Preservation rates | 8 weeks after chemoradiotherapy
  Sphincter Preservation rates 8 weeks post chemoradiotherapy at surgery.Percentage of patients who underwent sphincter salvage surgery after chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Tey, FRANZCR, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Ryan R, Gibbons D, Hyland JM, Treanor D, White A, Mulcahy HE, O'Donoghue DP, Moriarty M, Fennelly D, Sheahan K. Pathological response following long-course neoadjuvant chemoradiotherapy for locally advanced rectal cancer. Histopathology. 2005 Aug;47(2):141-6. doi: 10.1111/j.1365-2559.2005.02176.x. PMID 16045774